CLINICAL TRIAL: NCT06738316
Title: What is the Clinical Experience of Maintaining Patient Safety in Hospital in Patients With Temporary or Permanent Loss of Cognitive Function? A Mixed Methods Study
Brief Title: Clinical Experience of Maintaining Patient Safety in Hospital
Acronym: CEMPSIH
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 24065
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-11

CONDITIONS: Patient Safety
Keywords: Patient Safety; Fall prevention in hospitals; healthcare workers; simulation; focus group; critical decision method

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare Worker Focus Groups: Self nominated participants from various healthcare worker professions and jobs. Doctors, Nurses, Therapists and Support Staff
  Interventions: Behavioral: Simulation

INTERVENTIONS:
Behavioral: Simulation — Simulation of a patient safety incident in practice. The simulation closely replicates the workplace experience.

SUMMARY:
The key purpose of the study is to establish what the barriers to preventing accidental falls in hospital are, what interventions are perceived to work best in preventing falls and what could help. The study will attempt to disprove the null hypothesis that "there is no universal clinical experience of accidental fall prevention in hospitals with patients who have impaired cognitive function".

To gather an evidence base for the co-created design and testing of fall prevention interventions as part of the longer term PhD project.This is a multi-centre qualitative study utilising a purposive sampling strategy. Healthcare workers directly involved in preventing falls in hospital will be invited to contribute to the study via an email from their ward manager or clinical lead. Participants will be asked to respond directly to the investigator to indicate their interest in the study. They will be selected to ensure both Medical and Surgical wards are represented. Overall aim will be for up to 16 participants from the nursing team, registered and unregistered, up to 8 therapist participants and up to 8 doctors.This will provide 2 nurses, 1 therapist, 1 doctor in each simulation. This will provide 4 datasets for analysis and this process will be repeated at up to 4 Hospitals to deliver up to 16 datasets. Each group will participate in a 30 minute simulation followed by a semi structured focus group where critical decision method will be used to extract themes and codes to inductively generate a questionnaire for a further study. Patient and Public Involvement (PPI) representatives will be consulted on the outcomes of the focus groups.

DETAILED DESCRIPTION:
The National Institute for Health and Care Excellence clinical guidance CG161 recommends that all patients admitted to hospital over the age of 65 and those with specific underlying conditions between the age of 50 and 64 are considered at high risk of falls and a documented falls risk assessment is undertaken on admission. However, whilst advising the use of an appropriate multifactorial risk assessment (MFA) NICE also acknowledges that there is no evidence of the efficacy of most falls prevention methods in hospital and that high quality randomised controlled trials (RCT) conducted in the UK are required to improve the existing evidence base.

Falls are referred to as accidents but statistically they have been shown not to demonstrate a pattern of chance which suggests a causal process. Contributing factors leading to falls have been recognised as; postural stability, gait, sensory deficit, neuromuscular impairment, psychological conditions, impact of medications, environmental risks and medical risks such as stroke and cardiac issues. Significant research has been undertaken in relation to falls in the community and as such there are useful clinical guidelines published by both NICE and World Falls Guidelines for preventing and managing patients falls in their home. Whilst patients may be at less risk in their own environment, when admitted to hospital usually single or multiple risk factors apply, even if only for a limited period due to the nature of their presenting condition. It is therefore necessary to assess all patients who are admitted to hospital to establish the level of risk they face and to prescribe interventions with the goal of preventing an accidental fall.

In the UK, 30 - 50% of accidental falls in hospital lead to some injury and 1-3% of those sustain a fracture. In-patient falls are a significant cause of morbidity and mortality, with an estimated 247,000 occurring annually at a cost of £2.3billion to the NHS. In-patient falls have consistently been the biggest single category of reported incidents since the 1940's. Little has changed in the 39 years since the that paper and with falls accounting for 85% of all hospital acquired conditions in the USA it is safe to say this is a global issue. A recent Australian study estimated that the annual cost of attempts to prevent in-hospital falls across six health services consumed AU$590 million per year in resources. The areas of greatest investment were 18% physiotherapy, 14% 24 hour observation, 12% falls assessments and 11% falls prevention alarms and there is a lack of quality research to support their efficacy as falls prevention strategies. The generalisable level of success of these strategies is still not known. It seems that health services across the world are investing time and effort in strategies for which there is an absence of evidence. The recently published World Guidelines for Falls Prevention has confirmed there remains no research supporting the use of technology such as falls alarms or nonslip socks (NSS) in hospitals and as such recommends only standard falls prevention methods. As a result of increasing reimbursement costs for hospital treatments, in 2008 the Centres for Medicaid & Medicare Services, health insurance companies in the United States of America (US), removed reimbursement to hospitals for costs incurred by patient falls and any associated trauma resulting in increasing financial burden to hospitals. The impact on staff suffering 'second victim phenomena' as a result of adverse incidents and the cost to patients who suffer pain, disability, and death is incalculable.

ELIGIBILITY:
Inclusion Criteria:

* Any healthcare professional or associated support staff involved in the fall risk assessment of patients on admission to a standard care ward environment in hospital
* Any healthcare professional or associated support staff involved in the multifactorial assessment of patients in an acute ward environment
* Any healthcare professional or associated support staff involved in putting fall prevention measures in place in an acute ward environment
* Any healthcare professional or associated support staff involved in caring for patients and their relatives after an accidental fall in an acute ward environment
* Ability to give informed consent

Exclusion Criteria:

* Any healthcare worker with no medical or surgical ward experience
* Any healthcare worker under the age of 18 years old
* Any healthcare worker working exclusively in Critical Care or high dependency units or Paediatrics as countermeasures and levels of observation are different in these areas and have separate guidance and policies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals involved in the management or care of patients who are at risk of accidental falls in hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
To disprove the null hypothesis that "there is no universal clinical experience of accidental fall prevention in hospitals with patients who have impaired cognitive function". | September 2025
  Up to 32 multidisciplinary participants in each of 3 NHS Trusts will take part in a simulation of a ward based patient safety incident. They will then debate how closely this resembles their lived experience of managing patient safety in a ward environment. From this themes and codes will be analysed and the outcomes tested via questionnaire feedback from a larger broader population of healthcare workers. the questionnaire will be distributed to 4000 healthcare workers across the country. Statistical analysis of both quantitative and qualitative data will disprove or prove the null hypothesis.

SECONDARY OUTCOMES:
To inductively generate a questionnaire to be distributed to healthcare professionals and care workers in a future study. | September 2025
  Themes and codes will be analysed and the outcomes tested via questionnaire feedback from a larger broader population of healthcare workers. the questionnaire will be distributed to 4000 healthcare workers across the country. Statistical analysis of both quantitative and qualitative data will disprove or prove the null hypothesis.
To gather an evidence base for the co-created design and testing of fall prevention interventions as part of the longer term PhD project | April 2026
  To generate a cross NHS Trust research group of up to 8 participants that will work collaboratively to co-create interventional clinical trials that will result in a reduction in falls/1000 bed days for each unit in which the design is tested. Additional performance measures will be reported to demonstrate the importance of context such as number of admissions, discharges, high dependency patients and length of stay. Qualitative data will be collected to establish acceptability of the intervention to healthcare workers.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - University Hospitals of Leicester, Leicester
  - Nottingham University Hospitals, Nottingham
  - Northern Care Alliance, Rochdale Care Organisation, Salford

IPD SHARING:
Plan to Share IPD: Undecided
The work is a collective experience and knowledge base. Any individual opinion will be shared within the focus group and a group perspective will be reported therefore individual participant data would be incomplete and therefore worthless. Demographics would not be relevant due to very small sample size.
  This will however be reconsidered once the questionnaire is designed and amended accordingly